CLINICAL TRIAL: NCT00768833
Title: Nasopharyngeal Carriage in Children After Introduction of General Pneumococcal Immunization in Germany
Brief Title: Study Evaluating the Nasopharyngeal Carriage in Healthy Children
Acronym: Carriage
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: 0887X1-4453
Record Dates: First submitted 2008-10-07; First posted 2008-10-08 (Estimated); Last update posted 2014-08-21 (Estimated); Status verified 2014-08

CONDITIONS: Healthy Subjects
Keywords: S.pneumoniae healthy subjects; Healthy subjects

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to assess the prevalence of pneumococcal stereotypes in the nasopharynx of healthy children and to describe the changes of nasopharyngeal carriage at different ages over time.

ELIGIBILITY:
Inclusion Criteria:

Main inclusion criteria:

* Age at enrolment 3 to 4 month Main

Exclusion Criteria:

* Malformation or injury of the nasopharynx
* Known or suspected immunodeficiency
* Relevant immunosuppression
* Use of antibiotics up to 10 days prior to study inclusion

Ages: 3 Months to 4 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: community sample
Sampling Method: Non-Probability Sample
Enrollment: 242 (Actual)
Dates: Start 2008-10; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Number and frequency of S. pneumonia positive serotypes | 57 months

SECONDARY OUTCOMES:
Changes in number and frequency of S. pneumonia positive children at different ages over time | 57 month

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Offenbach, Germany

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=0887X1-4453&StudyName=Study%20Evaluating%20the%20Nasopharyngeal%20Carriage%20in%20Healthy%20Children